CLINICAL TRIAL: NCT06058481
Title: Comparing the Clinical Performance of BlockBuster vs Proseal-LMA in Unparalysed Patients Undergoing General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FF-2019-365; Fundamental data (Other: Universiti Kebangsaan Malaysia, Malaysia)
Record Dates: First submitted 2023-09-12; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Supraglottic Airway Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The investigator inserted the BlockBuster (supraglottic airway device) in Group A patients after induction of anaesthesia.
  Interventions: Device: Blockbuster
- Group B (Active Comparator): The investigator inserted the Proseal-LMA (supraglottic airway device) in Group B patients after induction of anaesthesia.
  Interventions: Device: Proseal-LMA

INTERVENTIONS:
Device: Blockbuster — The investigator inserted the BlockBuster in Group A patients.
  Arms: Group A
Device: Proseal-LMA — The investigator inserted the Proseal-LMA in Group B patients.
  Arms: Group B

SUMMARY:
Patients aged 19 to 78 years with ASA status I-II scheduled for elective surgery under general anesthesia, were recruited and randomized into two groups, Group A (BlockBuster) and Group B (Proseal-LMA). Anesthesia induction for both groups was standardized with no paralysis given. Supraglottic airway (SGA) insertion (either Blockbuster or Proseal-LMA) was executed by a single experienced investigator. The investigator inserted the BlockBuster in Group A patients and the Proseal-LMA in Group B patients. These parameters were compared between the groups; the number of attempts, time taken to achieve successful insertion, oropharyngeal leak pressure (OLP), fiberoptic view of SGA position, hemodynamics changes and complications from the insertion.

DETAILED DESCRIPTION:
This prospective, randomised single-blinded study, was conducted at the operation theatre of Universiti Kebangsaan Malaysia Medical Centre (UKMMC), following approval from the Institutional Ethics Committee of Universiti Kebangsaan Malaysia (UKM). The recruited patients were within the age range of 19 to 78 years, classified as American Society of Anesthesiologists Physical Status (ASA) class I or II, and underwent elective surgery under general anesthesia that required supraglottic airway (SGA) insertion. Exclusion criteria included a body mass index (BMI) over 35 kg/m2, limited mouth opening of less than two finger breath of inter-dental gap, edentulous, loose teeth, airway abnormalities, risk of aspiration, and known allergies to fentanyl and propofol.

During the pre-operative visit, patients were briefed about the study, and written informed consent was obtained. All recruited patients were fasted for at least 6 hours before the scheduled operation. No premedication was administered. Patients were then randomly assigned to either Group A (Blockbuster) or Group B (Proseal-LMA) using simple randomisation. SGA insertion was performed by a single operator with more than five years of experience using the Proseal-LMA and had received training using Blockbuster on a mannequin and successfully inserted it in 20 patients .

In the operation theatre, minimal standard monitoring was applied and followed by preoxygenation for three minutes. Anesthesia induction was conducted using intravenous (IV) fentanyl of 2 mcg/kg and IV propofol of 2 to 2.5 mg/kg. Additional propofol boluses of 10 to 20 mg were administered if anesthesia was inadequate and the doses were documented. Neuromuscular relaxant was not used. After achieving unconsciousness, mask ventilation was initiated with an oxygen and sevoflurane mixture until a Minimum Alveolar Concentration (MAC) of 1.3 was achieved. The depth of anesthesia was assessed by pupillary size and jaw relaxation prior to SGA insertion. The appropriate size of the SGA was chosen based on the manufacturer's recommendation according to the patient's body weight. Before SGA insertion, lubrication was applied to the outer cuff with a water-based lubricant and the cuff was fully deflated.

An assigned assistant recorded the number of attempts and time taken for successful insertion. The time taken for SGA insertion was measured from the moment SGA passes the patient's front incisor until the appearance of the first end-tidal CO2 (ETCO2) waveform on the capnography. The measurement of time was stopped and reset for subsequent attempts. The investigator inserted the BlockBuster in Group A patients and the Proseal-LMA in Group B patients. The Proseal-LMA is a reusable device and the items that used in this study was used less than 10 times previously. After SGA insertion, the cuff was inflated to a pressure of 60 cmH2O using a cuff pressure manometer. Successful insertion was determined by these three findings: chest expansion, no audible leak detected during manual bagging and the appearance of square wave capnograph tracing with ventilation generating expiratory tidal volumes of 6 to 8 ml/kg with an oxygen flow of 6 litre/min, adjustable pressure-limiting (APL) valve closed at 30 cmH2O. An audible leak was determined by listening at the mouth or lateral thyroid cartilage using a stethoscope for audible noise.

Following successful SGA insertion, a gastric tube sized 12 or 14 Fr was inserted. Oropharyngeal leak pressure (OLP) was assessed by setting the APL valve of the circle system at 30 cmH2O with a fresh gas flow of 3L/min. The OLP was determined by observing the airway pressure at equilibrium until an audible noise was heard over the mouth with a stethoscope. For safety reasons, the OLP was kept below 40 cmH2O and pressure was recorded.

The removal of SGA from the oral cavity was considered a failed attempt. If there was a failure of insertion or failure of placement of SGA (inadequate chest expansion, inability to generate adequate tidal volume or audible leak), the patient was ventilated again with 100% oxygen and 3% sevoflurane to maintain SpO2 above 95% before the next attempt. If inappropriate SGA size due to a large leak (small size) or difficult insertion (large size), new SGA insertion with different sizes was allowed once in this study. A maximum of three attempts was allowed, after which the patient was considered as failed SGA insertion. The subsequent airway management was determined by the responsible anaesthesiologist. The patient was dropped out of this study and excluded from the analysis if failed SGA insertion after three attempts and surgery duration exceeding two hours.

Anesthesia was maintained with sevoflurane in an air-oxygen mixture and ventilation was adjusted to achieve an adequate tidal volume of 6 to 8 ml/kg. Blood pressure, mean arterial pressure (MAP), heart rate (HR), ETCO2 and saturation were recorded at pre-induction, during induction, as well as at 5 and 10 minutes after SGA insertion. The position of SGA after insertion in relation to the laryngeal inlet was verified using an intubating bronchoscope Ambu aScope 4 Broncho Regular Endoscope (Ambu A/S, Denmark) with a working channel width of 2.2mm. The laryngeal view obtained was scored according to Keller et al. grading system: Grade 4, only vocal cords visible; Grade 3, vocal cords plus posterior epiglottis visible; Grade 2, vocal cords plus anterior epiglottis visible; Grade 1, vocal cords not visible.

The presence of airway complications related to SGA insertion such as laryngospasm, bronchospasm, gagging, coughing and aspiration was recorded and managed by the responsible anaesthesiologist. At the end of the operation, sevoflurane was discontinued, and the patient was allowed to breathe spontaneously in 100% oxygen. The SGA was removed once the patient had regained consciousness, was responsive to verbal commands and was able to breathe spontaneously generating tidal volumes of at least 6 to 8 ml/kg. Following SGA removal, the device was checked for blood-stained secretion and documented. The duration of anesthesia was recorded and was defined as the time taken from anesthesia induction until SGA removal. Patients were evaluated for the incidence of sore throat in the recovery area and at 24 hours post-anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* age range of 19 to 78 years
* classified as American Society of Anesthesiologists Physical Status (ASA) class I or II
* underwent elective surgery under general anesthesia that required supraglottic airway insertion.

Exclusion Criteria:

* patients with a body mass index (BMI) over 35 kg/m2.
* patients with limited mouth opening of less than two finger breath of inter-dental gap, edentulous, loose teeth and airway abnormalities.
* patients who at risk of aspiration.
* patients with known allergies to fentanyl and propofol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure measurement to assess efficacy of airway seal by the supraglottic airway device | 1 year
  Oropharyngeal leak pressure (OLP) was assessed by setting the adjustable pressure-limiting (APL) valve of the circle system at 30 cmH2O with a fresh gas flow of 3L/min. The OLP was determined by observing the airway pressure at equilibrium until an audible noise was heard over the mouth with a stethoscope. The measurement unit is cmH2O. For safety reasons, the OLP was kept below 40 cmH2O.

SECONDARY OUTCOMES:
First pass success rate | 1 year
  Number of patients who successfully being inserted with the supraglottic device on the first attempt
Number of supraglottic airway insertion attempt | 1 year
  Number of supraglottic airway insertion attempt in each patients
Supraglottic airway insertion time | 1 year
  Supraglottic airway (SGA) insertion time was measured from the moment SGA passes the patient's front incisor until the appearance of the first end-tidal CO2 waveform on the capnography. The measurement unit is seconds.

OTHER OUTCOMES:
Position of supraglottic airway device after insertion | 1 year
  The position of supraglottic airway in relation to the laryngeal inlet was verified using an intubating bronchoscope Ambu aScope 4 Broncho Regular Endoscope (Ambu A/S, Denmark) with a working channel width of 2.2mm. The laryngeal view obtained was scored according to Keller et al. grading system: Grade 4, only vocal cords visible; Grade 3, vocal cords plus posterior epiglottis visible; Grade 2, vocal cords plus anterior epiglottis visible; Grade 1, vocal cords not visible.
Mean arterial pressure during supraglottic airway insertion | 1 year
  Mean arterial pressures (in mmHg) were recorded at pre-induction, during induction, as well as at 5 and 10 minutes after supraglottic airway insertion.
Heart rate during supraglottic airway insertion | 1 year
  Heart rates (in beats per minute) were recorded at pre-induction, during induction, as well as at 5 and 10 minutes after supraglottic airway insertion.
Airway complications related to supraglottic airway insertion | 1 year
  The presence of airway complications related to supraglottic airway insertion such as laryngospasm, bronchospasm, gagging, coughing and aspiration was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Budiman, M.D., Principal Investigator — Faculty of Medicine, Universiti Kebangsaan Malaysia
Locations (1):
- Hospital Canselor Tuanku Muhriz Universiti Kebangsaan Malaysia, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No